CLINICAL TRIAL: NCT05068622
Title: Role of the Gastric Tube in the Preoperative Management of Hypertrophic Pyloric Stenosis
Brief Title: Gastric Tube in Pyloric Stenosis
Acronym: SONPYL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0188
Record Dates: First submitted 2021-09-15; First posted 2021-10-06 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Hypertrophic Pyloric Stenosis; Respiratory Complication
Keywords: Hypertrophic Pyloric Stenosis; gastric tube; Respiratory Complication
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with nasogastric tube before surgery
- patients without nasogastric tube before surgery

SUMMARY:
Pyloric stenosis is a current condition in pediatric surgery. The medical management prior to surgery consists of ionic correction. The nasogastric tube is commonly used to prevent gastric fluid inhalation before surgery, but there is no study on it benefits in this specific use. Other studies suggest that utilization of a gastric tube in pyloric stenosis may increase the duration of the medical treatment. The aim of the study is to evaluate the benefit of the nasogastric tube to prevent respiratory complications. This retrospective, monocentric and descriptive study include all patients hospitalized for pyloric stenosis in the university hospital in Amiens between 2014 and 2021. Patients with and without nasogastric tube prior to surgery are compared, regarding respiratory complications define as use of antibiotic, or oxygen therapy or infection in the lungs X-ray before surgery. The investigators analyze pre-operative data: vomiting, dehydration, time to ionic disorders correction and pain, and also notice the length of hospital stay. Data during hospitalization are analyzed and will be noticed the last medical contact represent by the post-operative consultation.

ELIGIBILITY:
Inclusion Criteria:

* all patients with hypertrophic pyloric stenosis

Exclusion Criteria:

* refusal of data collection and use from patient's parent or family

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all patients hospitalized for pyloric stenosis in the university hospital in Amiens between 2014 and 2021
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
occurrence of respiratory complications before surgery | baseline, pre-surgery
  respiratory complications are defined by antibiotic use and/or oxygenotherapy and/or infection in the lungs X-ray before surgery

SECONDARY OUTCOMES:
number of : pre-operative vomiting | baseline, pre-surgery
pre-operative comfort | baseline, pre-surgery
  pre-operative comfort is evaluated by the EDIN scale
pre-operative dehydration | baseline, pre-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Nord, Amiens, France

IPD SHARING:
Plan to Share IPD: No